CLINICAL TRIAL: NCT05597020
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, 2-way Cross-over Post Approval Study to Investigate the Efficacy of Daridorexant in Subjects With Insomnia and Comorbid Nocturia
Brief Title: A Study to Find Out if Daridorexant is Safe and Efficacious in Patients With Insomnia and Comorbid Nocturia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078A401; 2022-501246-30-00 (Other: EU CT Number)
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Insomnia Disorder; Nocturia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Nocturia | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: This is a multi-center, double-blind, randomized, placebo-controlled, 2-way cross-over post-approval study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 50 mg daridorexant (Experimental): Daridorexant will be taken orally, once daily in the evening within approximately 30 min before going to bed.
  Interventions: Drug: Daridorexant
- Placebo (Placebo Comparator): Matching placebo will be taken orally, once daily in the evening within approximately 30 min before going to bed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daridorexant — Daridorexant is available as oral film-coated tablets at a strength of 50 mg.
  Arms: 50 mg daridorexant
Drug: Placebo — Placebo matching daridorexant is provided as identical-looking oral tablets, formulated with the same inactive ingredients (excipients) as the active tablets.
  Arms: Placebo

SUMMARY:
A study to find out if daridorexant is safe and efficacious in patients with insomnia and comorbid nocturia

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (ICF) prior to any study-mandated procedure.
* Male or female subjects ≥ 55 years old at the time of signing the ICF.
* Insomnia complaints for at least 3 months prior to Visit 1.
* Insomnia Severity Index© (ISI©) score ≥ 13 at Visit 1.
* Nocturia severity: on average ≥ 3 nocturnal voids per night reported by the subjects for at least 1 month prior to Visit 1.
* Ability to communicate well with the investigator, to understand the study requirements and judged by the investigator to be alert and oriented to person, place, time, and situation.

Exclusion Criteria:

* Woman of childbearing potential, pregnant or plans to become pregnant.
* Planned travel across ≥ 3 time zones during study.
* Life time history of suicidality assessed via Columbia Suicide Severity Rating Scale© (C-SSRS©).
* Regular caffeine consumption after 4 pm.
* Unable to refrain from smoking during the night.
* Known and documented diagnosis of narcolepsy, periodic limb movement disorder, moderate to severe obstructive sleep apnea, restless legs syndrome, circadian rhythm sleep-wake disorder, or rapid eye movement (REM) sleep behavior disorder.
* Known and documented diagnosis of Type 1 diabetes mellitus, uncontrolled Type 2 diabetes mellitus, central or nephrogenic diabetes insipidus, and primary/secondary polydipsia.
* Known and documented nocturia linked to urinary tract infection, neoplasms of bladder, prostate or urethral cancer, bladder or urethral calculi, or neurogenic voiding dysfunction within the last 6 months prior to Visit 1.
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of the results, such as drug or alcohol dependence or psychiatric disease.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (16):
- United States (5):
  - Quantum Clinical Trials, Miami Beach, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Ochsner LSU Health Shreveport-Regional Urology, Shreveport, Louisiana
  - Accellacare Research of Cary, Cary, North Carolina
- Germany (3):
  - Praxisklinik am Franziskushospital - Urologisches Zentrum Euregio, Aachen
  - ASR Advanced Sleep Research GmBH, Berlin
  - SOMNIBENE Institut für Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - UROCLINICA Barcelona, Barcelona
  - Hospital Universitario Puerta del Mar (HUPM), Cadiz
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospitalario Universitario de Canarias, San Cristóbal de La Laguna

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 sites in 3 countries (USA, Spain and Germany) screened 149 subjects, and 9 sites enrolled (i.e., randomized) at least one subject. Screening started on 18 January 2023 (first subject first visit) and the first subject was enrolled on 16 February 2023.
Pre-assignment Details: This study included a screening period of 14-21 days. Subjects who met the inclusion criteria and none of the exclusion criteria were eligible to be enrolled in the study and randomized to one of the two treatment sequences.
Groups:
- Daridorexant 50 mg, Then Placebo: Subjects first received a daridorexant 50 mg film-coated tablet once daily in the evening within approximately 30 min before going to bed, for 29 (± 2) days.
  After a washout period of 14 to 21 days, they then received a placebo film-coated tablet (matching daridorexant 50 mg) once daily in the evening within approximately 30 min before going to bed, for 29 (± 2) days.
- Placebo, Then Daridorexant 50 mg: Subjects first received a placebo film-coated tablet (matching daridorexant 50 mg) once daily in the evening within approximately 30 min before going to bed, for 29 (± 2) days.
  After a washout period of 14 to 21 days, they then received a daridorexant 50 mg film-coated tablet once daily in the evening within approximately 30 min before going to bed, for 29 (± 2) days.
Period: Treatment Period I
Arm/Group | Daridorexant 50 mg, Then Placebo | Placebo, Then Daridorexant 50 mg
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Washout
Arm/Group | Daridorexant 50 mg, Then Placebo | Placebo, Then Daridorexant 50 mg
Started | 30 | 30
Completed | 28 | 30
Not Completed | 2 | 0
Not completed — Forbidden medication | 2 | 0
Period: Treatment Period II
Arm/Group | Daridorexant 50 mg, Then Placebo | Placebo, Then Daridorexant 50 mg
Started | 28 | 30
Completed | 26 | 29
Not Completed | 2 | 1
Not completed — Advice from primary care physician | 1 | 0
Not completed — Subject lost investigational product | 1 | 0
Not completed — Private reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daridorexant 50 mg, Then Placebo | Placebo, Then Daridorexant 50 mg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Full Range); unit: years] | 63 [55 to 81] | 63 [55 to 80] | 63 [55 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 18 | 13 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 22 | 20 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
  Germany | 7 | 6 | 13
  Spain | 3 | 2 | 5
Subjective total sleep time (sTST) [Mean (Standard Deviation); unit: minutes] | 367.20 (58.60) | 353.17 (54.85) | 360.31 (56.72)
Number of nocturnal voids [Mean (Standard Deviation); unit: Number of nocturnal voids] | 3.74 (1.05) | 3.52 (0.89) | 3.63 (0.97)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in sTST
Description: Subjective total sleep time (sTST) is the total sleep time reported by the subject in the sleep diary questionnaire. A positive change from baseline indicates an increase in sTST.
  Baseline is the mean value based on the subject's sleep diary entries for sTST on the 7 days preceding randomization.
  Week 4 is the mean value based on the subject's sleep diary entries for sTST on study days 23-29 of each treatment period, regardless of premature treatment discontinuations (treatment policy strategy).
Time Frame: From baseline to Week 4 per treatment period.
Population: The analysis included all randomized subjects who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Groups:
- Daridorexant 50 mg: Subjects received a daridorexant 50 mg film-coated tablet once daily in the evening within approximately 30 min before going to bed, for 29 (± 2) days, in either crossover treatment period.
- Placebo: Subjects received a placebo film-coated tablet (matching daridorexant 50 mg) once daily in the evening within approximately 30 min before going to bed, for 29 (± 2) days, in either crossover treatment period.
Arm/Group | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 60 | 60
minutes | 56.6 [46.0 to 67.2] | 35.7 [25.0 to 46.4]
Statistical Analysis 1: Comparison: Daridorexant 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis; Treatment, period, week within period, and interaction of treatment and week were factors; baseline sTST assessment was covariate; Least Square mean difference vs placebo = 20.9, 95% CI 2-sided [8.0 to 33.7]

2. Other Pre Specified Outcome: Change From Baseline to Week 4 in Number of Nocturnal Voids Assessed Using a Voiding Diary
Description: The number of nocturnal voids is the total of all nocturnal voids reported by the subject in the voiding diary.
  Baseline is the mean value based on subject's voiding diary entries for number of nocturnal voids across 3 nights during the screening period.
  Week 4 is the mean value based on subject's voiding diary entries for number of nocturnal voids across the 3 nights immediately preceding the Week 4 visit of each treatment period, regardless of premature treatment discontinuations (treatment policy strategy).
Time Frame: From baseline to Week 4 per treatment period.
Population: The analysis included all randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: number of nocturnal voids
Arm/Group | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 60 | 60
number of nocturnal voids | -1.6 (1.4) | -1.3 (1.3)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events from the 29-day (± 2 days) treatment periods are reported. Adverse events were considered treatment-emergent if the date of onset or worsening was from the first intake of study treatment up to 5 days after the end of study treatment.
Arm/Group | Daridorexant 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 6/60 | 2/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant 50 mg (N=60) | Placebo (N=58)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 3 (3) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to the sponsor for review at least 60 days prior to submission for publication or presentation at a congress. Upon review, the sponsor may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator is permitted to write a publication during such a review period.

DOCUMENTS (2):
  • Study Protocol (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT05597020/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT05597020/SAP_001.pdf